CLINICAL TRIAL: NCT02733822
Title: A Pilot, Phase 1, Open-Labelled, 4 Period, Randomised, Crossover Study to Evaluate the Pharmacokinetics of Naloxone When Given by the IV, IM and Buccal Routes of Administration in Healthy Male Subjects
Brief Title: Buccal Versus Injectable Naloxone: a Phase I Healthy Volunteer Study
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: KCL/NALOX/01/14
Record Dates: First submitted 2016-03-08; First posted 2016-04-12 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Drug Overdose; Opioid-Related Disorders
Keywords: opiate; heroin; opioid; overdose; naloxone
MeSH Terms: conditions — Drug Overdose; Opioid-Related Disorders | interventions — Naloxone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- IMP: buccal naloxone (single dose) (Experimental): 0.8 mg buccal (solution) of 1 mg/ml Naloxone Hydrochloride Injection
  Interventions: Drug: Naloxone
- IMP: buccal naloxone (double dose) (Experimental): 1.6 mg buccal (solution) of 1 mg/ml Naloxone Hydrochloride Injection
  Interventions: Drug: Naloxone
- Intramuscular (IM) reference (Active Comparator): 0.8 mg IM injection of 1 mg/ml Naloxone Hydrochloride Injection
  Interventions: Drug: Naloxone
- Intravenous (IV) reference (Active Comparator): 0.8 mg IV injection of 1 mg/ml Naloxone Hydrochloride Injection
  Interventions: Drug: Naloxone

INTERVENTIONS:
Drug: Naloxone
  Other Names: naloxone-hydrochloride

SUMMARY:
Naloxone is the standard treatment in response to cases of suspected opiate overdose.

Buccal formulation of naloxone is a novel alternative to the licensed naloxone injection which, by removing the risk of accidental needle-stick, may be safer and easier to administer.

Current UK policy allows the emergency administration of naloxone by any member of the general public (Strang, Kelleher, Best, Mayet, & Manning, 2006), and the preventative provision of naloxone to drug users and their family members ("take-home naloxone") is possible on a prescription basis. Thus, buccal naloxone may be particularly suitable for administration by family members who are providing interim overdose management care while awaiting the arrival of an ambulance.

The aim of this study is to examine the bioavailability and dose proportionality of buccal naloxone compared with the licensed injection standards (intravenous, intramuscular).

The investigators hypothesise that buccal naloxone is not inferior to the injection reference in absorption kinetics, i.e. time elapsed till peak concentration (Tmax; primary outcome), peak plasma concentration (Cmax), overall absorption (AUC), bioavailability (F%) and, duration of action (mean terminal half-life; T1/2).

The investigators propose a pharmacokinetic pilot investigation with within-subjects (crossover) design, comparing two doses (0.8 mg; 1.6 mg) of buccal naloxone hydrochloride solution to the licensed intramuscular (IM; 0.8 mg) and intravenous (IV; 0.8 mg) routes of injection. The investigators will invite four healthy (i.e., non-opioid using) male volunteers (n=4, not powered), each of whom will attend four experimental sessions at counterbalanced sequence. Each volunteer will receive naloxone hydrochloride doses of 0.8 mg IM, 0.8 mg IV, 0.8 mg buccal, and 1.6 mg buccal, with only one dose administered per session.

Blood concentrations will be measured at selected times during each session to establish speed of naloxone absorption, time to peak concentration, estimated half-life, and overall bioavailability. This dose-ranging pilot will inform future work by providing preliminary data on buccal naloxone absorption into the bloodstream and by establishing feasibility of the buccal route for naloxone delivery.

DETAILED DESCRIPTION:
Blood samples (3 ml) will be collected at -5, +1, 2, 3, 4, 6, 8, 10, 12.5, 15, 30, 45, 60, 75, 90, 120, 150, 180, 240, 300, 360, 420, and 480 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. Adult males aged 18 to 64 years inclusive and between 19 and 29.9 kg/m2 body mass index (BMI).
2. Subjects who are healthy as determined by pre-study medical history and physical examination.
3. Subjects who are able and willing to give written informed consent.
4. Medical history must be verified by either a personal physician or medical practitioner as appropriate.

Exclusion Criteria:

1. Subjects who do not conform to the above inclusion criteria.
2. Subjects who have a clinical condition (such as abnormal liver function, renal or cardiac issues) which, in the opinion of their personal physician or other examining medical practitioner, makes participation in the study inappropriate.
3. Subjects who have a clinically relevant surgical history.
4. Subjects who have a clinically relevant family history.
5. Subjects who have a history of relevant atopy.
6. Subjects who have a history of drug hypersensitivity relevant to naloxone.
7. Subjects who have a history of alcoholism.
8. Subjects who have a history of drug abuse.
9. Subjects who consume more than 42 units of alcohol a week. (unit = 1 glass of wine (125 mL) = 1 measure of spirits = ½ pint of beer)
10. Subjects who have an acute infection (such as influenza) or relevant lesion (such as oral tract) at the time of screening or admission. Subjects can be rescreened once they have recovered. At re-screening, a urine test of drugs of abuse and alcohol parameters will need to be repeated.
11. Subjects who have used prescription drugs within 4 weeks of first dosing.
12. Subjects who have used over the counter medications containing codeine or other opiates within 7 days of first dosing, unless agreed as not clinically relevant by the Principal Investigator. Details will be documented in source data.
13. Subjects who have used any investigational drug in any clinical trial within 3 months of receiving the last dose.
14. Subjects who have received the last dose of IMP greater than 3 months ago but who are on extended follow-up
15. Subjects who cannot communicate reliably with the Investigator.
16. Subjects who are unlikely to co-operate with the requirements of the study.

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Tmax | Within 8-hour sampling period
  Time elapsed till peak concentration

SECONDARY OUTCOMES:
Peak plasma concentration is assessed as Cmax | Within 8-hour sampling period
  Peak concentration
Absorption of the active ingredient is determined as Area under the Curve (AUC) | Within 8-hour sampling period
  Overall absorption (AUC = Area Under the Curve)
Absolute bioavailability of buccal naloxone relative to intravenous naloxone is assessed as F% | Within 8-hour sampling period
  Absolute bioavailability relative to the IV reference (dose-corrected AUC for non-intravenous Buccal AUC divided by intravenous AUC multiplied by 100
Mean terminal half-life is assessed for all participants as T1/2 | Within 8-hour sampling period
  mean terminal half-life

CONTACTS AND LOCATIONS:
Overall Officials: John Strang, MBBS, MD, Principal Investigator — King's College London

IPD SHARING:
Plan to Share IPD: Undecided
There is no plan to provide access to to raw data.